CLINICAL TRIAL: NCT03428035
Title: Neutral Formulated and Designed Package Insert or Only Verbal Information Compared to Package Insert According EU-directive: a Pilot Randomised Controlled Trial to Analyse the Influence on the Nocebo Effect and Non-adherence
Brief Title: The Impact of a Neutral Formulated and Designed Package Insert on Nocebo-effect.
Acronym: NEUPANO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Witten/Herdecke (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Tim Mathes, Dr. Tim Mathes, University of Witten/Herdecke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: V01-01
Record Dates: First submitted 2018-02-02; First posted 2018-02-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Orthopedic Surgery
Keywords: Randomized controlled trial; package insert; nocebo
MeSH Terms: interventions — Product Labeling; Patient Education as Topic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Modified Package Insert (Experimental): Simplified and focused on neutral risk perception. The representations and formulations are based on the findings from research on evidence-based patient information and risk communication. The package insert contains the same information as the statutory package insert to ensure that it complies with the legal requirements.
  Interventions: Other: Package Insert
- Verbal Information (No Intervention): The patient is informed verbally about side effects and does not receive any package insert.
- Control (Active Comparator): Package insert according to EU Directive 2001/83 / EC (usual package insert)
  Interventions: Other: Package Insert

INTERVENTIONS:
Other: Package Insert — Modified package insert of Ibuprofen given postprocedural as pain medication
  Other Names: Patient Education
  Arms: Control; Modified Package Insert

SUMMARY:
Background The nocebo effect describes the association between the expectation of negative effects, (e.g. side effects) and the actual occurrence of negative effects. Studies have shown that the nocebo effect can be influenced by (risk) communication. Till today there is no study that compares different types of information on adverse events regarding the strength of the nocebo effect.

Aim The aim of this pilot randomized controlled trial is to analyse the influence of different communication types on the frequency and intensity of adverse events and adherence. To increase the relevance and applicability of the results the study intervention builds up on package inserts because these are the most widespread form of information on side effects.

Methods Patients It is planned to include 60 patients in the study.

Intervention

* Modified package insert: simplified and focused on neutral risk perception. The representations and formulations are based on the findings from research on evidence-based patient information and risk communication. The package insert contains the same information as the statutory package insert to ensure that it complies with the legal requirements.
* Verbal information about side effects: The patient is informed verbally about side effects and does not receive any package insert.

Control Package insert according to EU (European Union) Directive 2001/83 / EC (European Commission) (usual package insert).

Outcomes

* Number of patient reported adverse events (primary outcome).
* Adherence (correct initiation of therapy, correct intake amount, premature discontinuation of therapy).
* Resource use (e.g. provider contacts).

Type of study Monocentric, outcome assessor, three-arm, randomised controlled pilot trial.

ELIGIBILITY:
Inclusion Criteria:

* elective orthopaedic surgery
* planned intake of ibuprofen 600 mg to treat postoperative pain
* postoperative pain medication other than Ibuprofen 600 (Opioids, Opiate, Paracetamol) no longer than 1-2 days postoperative (until discharge)
* at least 18 years
* able to speak German
* no cognitive deficits
* written informed consent

Exclusion Criteria:

* serious comorbidity
* pain medication prior to surgery
* other medication with similar side effects
* polytrauma
* planned inpatient rehabilitation > one week after hospital discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patient reported adverse events | 6-9 days after surgery
  Any reported adverse events

SECONDARY OUTCOMES:
Adherence | 6-9 days after surgery
  Correct initiation of therapy, correct intake amount, premature discontinuation of therapy
Resource use | 6-9 days after surgery
  e.g. provider contacts

CONTACTS AND LOCATIONS:
Overall Officials: Tim Mathes, Dr., Principal Investigator — Witten/Herdecke University
Locations (1):
- Clinic for orthopedics, trauma surgery and sports traumatology, hospital Cologne Merheim, Cologne, North-Rhine-Westfalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and clinical study report will be shared as supplement with the journal publication
Supporting Information: Study Protocol, CSR
Time Frame: 2019
Access Criteria: Will be published as electronic supplement with the journal publication

REFERENCES:
- [Derived] Prediger B, Meyer E, Buchter R, Mathes T. Nocebo effects of a simplified package leaflet compared to unstandardised oral information and a standard package leaflet: a pilot randomised controlled trial. Trials. 2019 Jul 26;20(1):458. doi: 10.1186/s13063-019-3565-3. PMID 31349865